CLINICAL TRIAL: NCT05420584
Title: Phase Ⅱ Clinical Trial of Neoadjuvant Arterial Embolization Chemotherapy Combined Immune Checkpoint Inhibitor for Locally Advanced Rectal Cancer: A Single Arm Prospective Sturdy
Brief Title: Neoadjuvant Arterial Embolization Chemotherapy Combined PD-1 Inhibitor for Locally Advanced Rectal Cancer
Acronym: NECI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K2022129
Record Dates: First submitted 2022-06-12; First posted 2022-06-15 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Rectal Neoplasms
MeSH Terms: conditions — Rectal Neoplasms | interventions — tislelizumab; XELOX

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental arm (Experimental)
  Interventions: Procedure: Arterial chemoembolization; Drug: Tislelizumab Injection; Drug: XELOX; Diagnostic Test: Pelvic MRI; Procedure: Laparoscopic radical resection of rectal cancer

INTERVENTIONS:
Procedure: Arterial chemoembolization — The blood supplying artery of the tumor is selected for drug injection with Oxaliplatin 85mg/m2 combined Raltitrexed 3mg/m2. After drug injection, gelatin sponge is used for embolization.
Drug: Tislelizumab Injection — Tislelizumab Injection 200mg i.v. q3w, A total of 3 cycles are administered.
Drug: XELOX — Capecitabine 1,000 mg/m2 bid, po, on days 1-14 Oxaliplatin: 130 mg/m2, i.v. day 1 Cycles are repeated on day 22. A total of 3 cycles are administered.
Diagnostic Test: Pelvic MRI — Pelvic MRI to evaluate efficacy
Procedure: Laparoscopic radical resection of rectal cancer — Surgical treatment for patients who meet the surgical conditions

SUMMARY:
Rectal cancer is one of the common malignant tumors of the digestive tract. Some patients with rectal cancer are already advanced tumors when they are first diagnosed. At this time, the tumor has local infiltration, the probability of recurrence and metastasis after surgical resection is high, and even radical tumor resection cannot be performed. Neoadjuvant chemotherapy and radiotherapy have become one of the important treatment methods for these patients to increase the rate of radical tumor resection. However, a series of side effects of neoadjuvant radiotherapy can even continue after the end of radiotherapy, and even increase the incidence of postoperative complications. Superselective arterial interventional chemotherapy has been widely used in preoperative neoadjuvant chemotherapy for various tumors, and its efficacy in rectal cancer has also been confirmed. In addition, as a hot spot in tumor treatment, tumor immunotherapy has shown exciting effects in the NICHE study of neoadjuvant immunotherapy before colon cancer surgery. Moreover, Oxaliplatin is a classic chemotherapeutic drug that induces Immunogenic cell death effects, which induce antitumor immunity.

Therefore, in order to optimize the preoperative neoadjuvant therapy plan, the investigators propose a treatment method of superselective arterial chemoembolization combined with immunotherapy and systemic chemotherapy, in order to obtain better preoperative conversion therapy effect and reduce the adverse reactions of neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed rectal adenocarcinoma (immunohistochemistry, polymerase chain reaction(PCR) or next-generation sequencing(NGS) sequencing methods are acceptable).
2. Magnetic resonance imaging (MRI) measurement of tumor inferior margin ≤12cm from the anus.
3. MRI staging is cT3-4 N0 or cT1-4 N+, no multiple primary cancers or distant metastasis.
4. Life expectancy ≥ 1 year.
5. No anti-tumor therapy, no contraindications to interventional embolization, immunotherapy and chemotherapy.
6. Patients who understand the study protocol and are willing to participate in this study provide written informed consent.

Exclusion Criteria:

1. Refuse to participate in this study.
2. Multifocal colorectal cancer.
3. Past history of malignancy, excluding basal cell carcinoma/papillary thyroid carcinoma/various types of carcinoma in situ.
4. Inability to receive chemotherapy, such as but not limited to bone marrow suppression, etc.
5. Major organ diseases (such as but not limited to chronic obstructive pulmonary disease, coronary heart disease and renal insufficiency, etc.) during acute exacerbation and or severe acute infectious diseases (such as but not limited to hepatitis, pneumonia and myocarditis, etc.), American Society of Anesthesiologists(ASA) score > 3.
6. Mental disability or illiteracy or language and communication barriers cannot understand the research protocol.
7. There are contraindications to arterial puncture, such as but not limited to severe arteriosclerosis or even atresia, coagulation dysfunction, long-term use of anticoagulants and cannot be stopped, etc.
8. Obstruction or high risk of obstruction by rectal tumor and/or bleeding and/or perforation.
9. Peripheral sensory nerve disorder, unable to receive oxaliplatin-based chemotherapy.
10. Lateral pelvic lymph node metastasis (mainly supplied by the internal iliac artery).
11. Pregnancy or breastfeeding.
12. Contraindications for MRI。
13. Consecutive use of corticosteroids for more than 3 days within 1 month before signing the consent form。
14. MRI assessment was T4b or MRF positive。
15. Other scenarios deemed inappropriate by the investigators for this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Imaging Tumor Regression Rate | From date of the start of drugs treatment until the end of drugs treatment (nearly 3 weeks)
  Tumor regression on imaging after neoadjuvant therapy

SECONDARY OUTCOMES:
Pathologic Complete Response | From date of the start of drugs treatment until the operation is completed (nearly 4 weeks)
  There is no histological evidence of malignancy in the primary tumor and metastatic regional lymph nodes, or there is only a carcinoma in situ component
Disease Free Survival | 36 months
  Time from postoperative disease-free survival to disease recurrence or metastasis
Safety (The side effects) | 36 months
  The side effects of this study
Pathological Tumor Regression Rate | From date of the start of drugs treatment until the end of drugs treatment (nearly 3 weeks)
  Tumor regression on pathology after neoadjuvant therapy

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Affiliated Hospital of Zhejiang University School of Medicine, Yiwu, Zhejiang, China

REFERENCES:
- [Background] Patel UB, Taylor F, Blomqvist L, George C, Evans H, Tekkis P, Quirke P, Sebag-Montefiore D, Moran B, Heald R, Guthrie A, Bees N, Swift I, Pennert K, Brown G. Magnetic resonance imaging-detected tumor response for locally advanced rectal cancer predicts survival outcomes: MERCURY experience. J Clin Oncol. 2011 Oct 1;29(28):3753-60. doi: 10.1200/JCO.2011.34.9068. Epub 2011 Aug 29. PMID 21876084
- [Result] Chalabi M, Fanchi LF, Dijkstra KK, Van den Berg JG, Aalbers AG, Sikorska K, Lopez-Yurda M, Grootscholten C, Beets GL, Snaebjornsson P, Maas M, Mertz M, Veninga V, Bounova G, Broeks A, Beets-Tan RG, de Wijkerslooth TR, van Lent AU, Marsman HA, Nuijten E, Kok NF, Kuiper M, Verbeek WH, Kok M, Van Leerdam ME, Schumacher TN, Voest EE, Haanen JB. Neoadjuvant immunotherapy leads to pathological responses in MMR-proficient and MMR-deficient early-stage colon cancers. Nat Med. 2020 Apr;26(4):566-576. doi: 10.1038/s41591-020-0805-8. Epub 2020 Apr 6. PMID 32251400
- [Derived] Fan Y, Zhu X, Xu C, Ding C, Hu J, Hong Q, Wang J. Neoadjuvant Arterial Embolization Chemotherapy Combined PD-1 Inhibitor for Locally Advanced Rectal Cancer (NECI Study): a protocol for a phase II study. BMJ Open. 2023 Mar 13;13(3):e069401. doi: 10.1136/bmjopen-2022-069401. PMID 36914193